CLINICAL TRIAL: NCT03234543
Title: Remote Ischemic Conditioning (RIC) to Decrease Post-Operative Complications After Major Abdominal Surgery - A Phase IIa Trial
Brief Title: Remote Ischemic Conditioning in Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Baburao Koneru, MD, MPH, Professor of Surgery, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro20160001420
Record Dates: First submitted 2017-07-25; First posted 2017-07-31 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Laparotomy; Laparoscopy; Retroperitoneal Disease; Pelvis Disease; Pancreatic Diseases; Liver Diseases; Gastrointestinal Disease; Urologic Diseases; Complication of Surgical Procedure
Keywords: Abdominal Surgery; Pre-conditioning; Remote Ischemic Conditioning; Post-Operative Complications; Acute Phase Response
MeSH Terms: conditions — Pancreatic Diseases; Liver Diseases; Gastrointestinal Diseases; Urologic Diseases; Acute-Phase Reaction

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, double - masked clinical trial of RIC will be conducted in adult patients undergoing major abdominal surgery at University Hospital in Newark, NJ. Participants will be randomized into two groups: RIC and No RIC.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study will be conducted in a double-masked fashion. Investigative team member/s that will carry out randomization and administer the intervention will not be involved in evaluation of clinical and laboratory outcomes. The primary surgical team, nurses, and any consulting services caring for the patient will be unaware of the group assignment. Other care providers will not be informed of the group assignment. Outcome assessors will not be involved in randomization and administration of the RIC intervention. Adequate steps are in place to mask the outcome assessors (clinical and laboratory) from knowing group assignment.
  Subjects will be masked from recognizing which group they are in in the following manner: a) Subjects will not be informed of the group assignment throughout their participation in the study; b) subjects randomized to No RIPC will have a tourniquet placed on the thigh and inflated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Conditioning (Experimental): The RIC intervention consists of 5 minutes of inflation of a pneumatic tourniquet placed mid-thigh followed by 5 minutes of deflation, repeated for 3 cycles. The pressure used will be 250 mmHg for the pre-operative intervention. Subsequent tourniquet pressures will be 50 mmHg above the patient's systolic blood pressure.
  Interventions: Procedure: Remote ischemic conditioning
- No Remote Ischemic Conditioning (Sham Comparator): The No RIC group will receive a sham intervention at all the same time points. The thigh tourniquet will be inflated to only 20 mmHg (to mask the intervention from the subject).
  Interventions: Procedure: No Remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Placement of blood pressure cuff to lower extremity in order to induce temporary and reversible ischemia.
  Arms: Remote Ischemic Conditioning
Procedure: No Remote ischemic conditioning — Placement of blood pressure cuff to lower extremity with minimal inflation without inducing ischemia.
  Arms: No Remote Ischemic Conditioning

SUMMARY:
This phase II randomized (1:1) controlled trial will examine the effects of remote ischemic conditioning (RIC) on the outcomes of major abdominal surgery. One hundred subjects will be enrolled at a single institution - University Hospital - Newark. The study population are patients undergoing major abdominal surgery (anticipated to be >/= 2 hrs long with a hospital stay >/= 2 days). Subjects in the treatment group will receive lower limb ischemic conditioning at 3 different time points: before surgery, POD 1 and POD 2. The primary outcome is the 30-day comprehensive complications index (CCI). Key secondary outcomes are changes in systemic inflammatory markers in peripheral blood and 30-day mortality.

DETAILED DESCRIPTION:
STUDY GOALS AND OBJECTIVES:

1. To obtain preliminary data regarding postoperative complications in subjects undergoing abdominal surgery and receiving remote limb ischemic or sham conditioning.
2. To test whether remote limb ischemic conditioning (RIC) decreases systemic inflammatory response in patients undergoing major abdominal surgery.

HYPOTHESiS:

The central hypothesis of the research is that pre- and post-operative RIC in patients undergoing major abdominal surgery would decrease the systemic inflammatory response to major abdominal surgery and decrease postoperative complications.

STUDY DESIGN:

A prospective, randomized, double - masked clinical trial of RIC will be conducted in adult patients undergoing major abdominal surgery at University Hospital in Newark, NJ. Participants will be randomized into two groups: RIC and No RIC. RIC will be induced at three time points - the first after anesthesia induction but before commencement of surgery, and the second and the third on post-operative days 1 and 2, respectively. The RIC intervention consists of 5 minutes of inflation of a pneumatic tourniquet placed mid-thigh followed by 5 minutes of deflation, repeated for 3 cycles. The pressure used will be 250 mmHg for the pre-operative intervention. Subsequent tourniquet pressures will be 50 mmHg above the patient's systolic blood pressure. The No RIC group will receive a sham intervention at all the same time points. The thigh tourniquet will be inflated to only 20 mmHg. A Doppler probe will be used to assess pedal arterial flow in both groups. Blood samples will be collected at baseline, 1hr after skin closure, and 1hr after interventions 2 and 3.

STUDY POPULATION:

Adults (> 18 years of age) of both sexes scheduled for elective major abdominal surgery at University Hospital will be considered for inclusion. Major abdominal surgery is defined as peritoneal, retroperitoneal and pelvic surgery expected to last >/= 120 minutes (from incision to closure) with an expected hospital stay >/= 2 days. A list of surgeries considered for inclusion is included as Appendix A. Additional operations will be considered for inclusion if the study team and primary surgical team both agree that the procedure is a major abdominal surgery and that the duration of surgery is likely to be > 2 hours.

RISKS AND BENEFITS

1. Risks to Subjects During inflation of the tourniquet in awake patients (post-op), there is a risk of pain secondary to tourniquet inflation. The investigators believe this risk is small, and if it occurs, the patient will have the option to discontinue the intervention.

   There is a theoretical risk of injury to the limb receiving the RIC stimulus. However, such occurrences have not been reported to date in other clinical studies.

   During collection of blood samples, there is a theoretical risk of bleeding from the venipuncture site; however this risk is no greater than routine blood draw. The amount of blood drawn for study purposes will be small (less than 50 mL total anticipated).
2. Benefits to Subjects The anticipated benefit to subjects is fewer complications after major abdominal surgery. However, no such benefit may accrue. In addition, the study is expected to provide valuable information regarding how RIC might modulate stress response to major surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (> 18 years of age)
2. Both genders
3. Undergoing major abdominal surgery as above
4. Elective surgeries
5. Both outpatients and in-hospital patients
6. Post-op length of stay expected to be at least 2 days by the primary surgical service

Exclusion Criteria:

1. Subjects with lower extremity paralysis
2. Lower extremity amputees
3. Known, documented peripheral arterial disease
4. Body mass index > 45
5. Pregnancy
6. Trauma patients
7. Organ transplant recipients
8. Prior major surgery during current hospitalization (for instance, a patient undergoing re-laparotomy for a complication from a previous procedure)
9. Patient taking sulfonylureas or nitrates prior to or during admission (listed in Appendix B)

   a. These subjects are excluded because sulfonylureas are shown to abrogate the RIC effect whereas nitrates are shown to mimic the RIC effect in animal models.
10. Non-elective surgeries (urgent or emergent surgeries)
11. General surgical procedures with no planned intra-abdominal component

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-08 (Actual); Primary Completion 2019-06-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index | 30 days after surgery
  The CCI, a validated and scaled score of all surgical complications (range 0 [no complications] to 100 [death]) will be computed for each subject using the publically available website, http://www.assessurgery.com/.

SECONDARY OUTCOMES:
Completion all three interventions | Up to 3 days
  Proportions of subjects completing all three research interventions
Hospital days | Up to 30 days
  Number of days to discharge from the hospital after surgery
30-day mortality | Up to 30 days
  Proportions of patients dying within 30 days after surgery
Plasma complement levels (C2, C4b, C5, C5a, and C5b-9) | Up to 3 days
  Measured at baseline, an hour after skin closure, completion of second and third research intervention
Plasma cytokines levels (TNF-a, IL - 1, 6, 8 and 10) | Up to 3 days
  Plasma cytokine levels at baseline, an hour after skin closure, completion of second and third research intervention
Plasma acute phase reactant proteins (CRP, alpha-1- acid glycoprotein, FGN, and haptoglobin) | Up to 3 days
  Measured at baseline, an hour after skin closure, completion of second and third research intervention
Peripheral blood leukocyte gene expression profiles determined by RNA sequencing. | Up to 3 days
  Measured at baseline, an hour after skin closure, completion of second and third research intervention

CONTACTS AND LOCATIONS:
Overall Officials: Baburao Koneru, MD, MPH, Principal Investigator — Rutgers-NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Lausevic Z, Lausevic M, Trbojevic-Stankovic J, Krstic S, Stojimirovic B. Predicting multiple organ failure in patients with severe trauma. Can J Surg. 2008 Apr;51(2):97-102. PMID 18377749
- [Background] Kvarnstrom AL, Sarbinowski RT, Bengtson JP, Jacobsson LM, Bengtsson AL. Complement activation and interleukin response in major abdominal surgery. Scand J Immunol. 2012 May;75(5):510-6. doi: 10.1111/j.1365-3083.2012.02672.x. PMID 22229650
- [Background] Kvarnstrom A, Sokolov A, Swartling T, Kurlberg G, Mollnes TE, Bengtsson A. Alternative pathway activation of complement in laparoscopic and open rectal surgery. Scand J Immunol. 2012 Jul;76(1):49-53. doi: 10.1111/j.1365-3083.2012.02702.x. PMID 22486843
- [Background] Birnbaum Y, Hale SL, Kloner RA. Ischemic preconditioning at a distance: reduction of myocardial infarct size by partial reduction of blood supply combined with rapid stimulation of the gastrocnemius muscle in the rabbit. Circulation. 1997 Sep 2;96(5):1641-6. doi: 10.1161/01.cir.96.5.1641. PMID 9315559
- [Background] Leung CH, Caldarone CA, Wang F, Venkateswaran S, Ailenberg M, Vadasz B, Wen XY, Rotstein OD. Remote Ischemic Conditioning Prevents Lung and Liver Injury After Hemorrhagic Shock/Resuscitation: Potential Role of a Humoral Plasma Factor. Ann Surg. 2015 Jun;261(6):1215-25. doi: 10.1097/SLA.0000000000000877. PMID 25185480
- [Background] Konstantinov IE, Arab S, Kharbanda RK, Li J, Cheung MM, Cherepanov V, Downey GP, Liu PP, Cukerman E, Coles JG, Redington AN. The remote ischemic preconditioning stimulus modifies inflammatory gene expression in humans. Physiol Genomics. 2004 Sep 16;19(1):143-50. doi: 10.1152/physiolgenomics.00046.2004. Epub 2004 Aug 10. PMID 15304621
- [Background] Pang T, Zhao Y, Zhang NR, Jin SQ, Pan SQ. Transient limb ischemia alters serum protein expression in healthy volunteers: complement C3 and vitronectin may be involved in organ protection induced by remote ischemic preconditioning. Oxid Med Cell Longev. 2013;2013:859056. doi: 10.1155/2013/859056. Epub 2013 Dec 2. PMID 24363825
- [Background] Hausenloy DJ, Yellon DM. Remote ischaemic preconditioning: underlying mechanisms and clinical application. Cardiovasc Res. 2008 Aug 1;79(3):377-86. doi: 10.1093/cvr/cvn114. Epub 2008 May 2. PMID 18456674
- [Background] Ali ZA, Callaghan CJ, Lim E, Ali AA, Nouraei SA, Akthar AM, Boyle JR, Varty K, Kharbanda RK, Dutka DP, Gaunt ME. Remote ischemic preconditioning reduces myocardial and renal injury after elective abdominal aortic aneurysm repair: a randomized controlled trial. Circulation. 2007 Sep 11;116(11 Suppl):I98-105. doi: 10.1161/circulationaha.106.679167. PMID 17846333
- [Background] Meng R, Asmaro K, Meng L, Liu Y, Ma C, Xi C, Li G, Ren C, Luo Y, Ling F, Jia J, Hua Y, Wang X, Ding Y, Lo EH, Ji X. Upper limb ischemic preconditioning prevents recurrent stroke in intracranial arterial stenosis. Neurology. 2012 Oct 30;79(18):1853-61. doi: 10.1212/WNL.0b013e318271f76a. Epub 2012 Oct 3. PMID 23035060
- [Background] Zarbock A, Schmidt C, Van Aken H, Wempe C, Martens S, Zahn PK, Wolf B, Goebel U, Schwer CI, Rosenberger P, Haeberle H, Gorlich D, Kellum JA, Meersch M; RenalRIPC Investigators. Effect of remote ischemic preconditioning on kidney injury among high-risk patients undergoing cardiac surgery: a randomized clinical trial. JAMA. 2015 Jun 2;313(21):2133-41. doi: 10.1001/jama.2015.4189. PMID 26024502
- [Background] Meybohm P, Bein B, Brosteanu O, Cremer J, Gruenewald M, Stoppe C, Coburn M, Schaelte G, Boning A, Niemann B, Roesner J, Kletzin F, Strouhal U, Reyher C, Laufenberg-Feldmann R, Ferner M, Brandes IF, Bauer M, Stehr SN, Kortgen A, Wittmann M, Baumgarten G, Meyer-Treschan T, Kienbaum P, Heringlake M, Schon J, Sander M, Treskatsch S, Smul T, Wolwender E, Schilling T, Fuernau G, Hasenclever D, Zacharowski K; RIPHeart Study Collaborators. A Multicenter Trial of Remote Ischemic Preconditioning for Heart Surgery. N Engl J Med. 2015 Oct 8;373(15):1397-407. doi: 10.1056/NEJMoa1413579. Epub 2015 Oct 5. PMID 26436208
- [Background] Hausenloy DJ, Candilio L, Evans R, Ariti C, Jenkins DP, Kolvekar S, Knight R, Kunst G, Laing C, Nicholas J, Pepper J, Robertson S, Xenou M, Clayton T, Yellon DM; ERICCA Trial Investigators. Remote Ischemic Preconditioning and Outcomes of Cardiac Surgery. N Engl J Med. 2015 Oct 8;373(15):1408-17. doi: 10.1056/NEJMoa1413534. Epub 2015 Oct 5. PMID 26436207
- [Background] Gonzalez NR, Hamilton R, Bilgin-Freiert A, Dusick J, Vespa P, Hu X, Asgari S. Cerebral hemodynamic and metabolic effects of remote ischemic preconditioning in patients with subarachnoid hemorrhage. Acta Neurochir Suppl. 2013;115:193-8. doi: 10.1007/978-3-7091-1192-5_36. PMID 22890668
- [Background] Li S, Ma C, Shao G, Esmail F, Hua Y, Jia L, Qin J, Ren C, Luo Y, Ding Y, Borlongan CV, Ji X. Safety and Feasibility of Remote Limb Ischemic Preconditioning in Patients With Unilateral Middle Cerebral Artery Stenosis and Healthy Volunteers. Cell Transplant. 2015;24(9):1901-11. doi: 10.3727/096368914X683520. Epub 2014 Jul 30. PMID 25198862
- [Background] Bilgin-Freiert A, Dusick JR, Stein NR, Etchepare M, Vespa P, Gonzalez NR. Muscle microdialysis to confirm sublethal ischemia in the induction of remote ischemic preconditioning. Transl Stroke Res. 2012 Jun;3(2):266-72. doi: 10.1007/s12975-012-0153-1. Epub 2012 Apr 10. PMID 24323782

DOCUMENTS (3):
  • Informed Consent Form (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT03234543/ICF_002.pdf
  • Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT03234543/SAP_003.pdf
  • Study Protocol (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT03234543/Prot_004.pdf